CLINICAL TRIAL: NCT02100709
Title: The Effect of BiLevel Pressure Support NonInvasive Ventilation on Quality of Life and Exercise Capacity in a COPD Exercise Rehabilitation Program
Brief Title: The Effect of NIV on QoL and Exercise Capacity in a COPD Exercise Rehabilitation Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sample size calculation would have been overinflated; re-think study design
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMD_NIV_COPD_001
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Control Arm (No Intervention): This arm will perform the pulmonary rehabilitation as specified with no respiratory assistance.
- Intervention Arm (Active Comparator): This arm will conduct the pulmonary rehabilitation program with BiLevel Noninvasive Ventilation assistance from a ResMed ventilator.
  Interventions: Device: BiLevel Noninvasive Ventilation

INTERVENTIONS:
Device: BiLevel Noninvasive Ventilation — Positive pressure applied through an oro-nasal mask. The pressure is altered between inspiration and expiration.
  Other Names: NIV; BiPAP; Pressure Support Ventilation; PSV
  Arms: Intervention Arm

SUMMARY:
This trial hopes to demonstrate the effect of 4 weeks of outpatient exercise rehabilitation on COPD patients. In particular the effect on:

* the amount of daily physical activity
* Quality of life
* The 6-minute walk distance
* Time to exacerbation

and compare it to the effect of 4 weeks of outpatients rehabilitation with Noninvasive Ventilation as an adjunct therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD III+IV
* Age >18 years
* Former NIV treatment for at least 6 weeks with a positive end-expiratory pressure of at least 4 cmH2O and a pressure support of 8 cmH2O or higher

Exclusion Criteria:

* Pulmonary Exacerbation requiring antibiotic treatment or hospitalization during the last 6 weeks
* non-pulmonary Exercise impairment (amputation, severe heart disease, etc)
* any disease that precludes exercise training
* inability to understand the patient information
* substance abuse
* oxygen requirement of more than 6l O2/min during exercise

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Daily Physical Activity | 3 Months
  The primary outcome will be measured by daily activity using accelerometer arm bands. This will be measured at the beginning of the rehabilitation program, at the end and at a 3 month follow up.
Exercise Capacity | 6 Weeks
  6 Minute Walking Distance will be measured every week during the exercise program.

SECONDARY OUTCOMES:
Quality of Life | 3 Months
  Using the St. George Respiratory Questionnaire before and after rehabilitation, quality of life will be measured.
Dyspnoea | 6 Weeks
  Change in Dyspnoea after end of exercise will be assessed using the Multidimensional Dyspnoea Profile and the BORG scale.
Change in Physiological Parameters | 3 Months
  Maximum training intensity, body weight and muscle diameter will be tracked throughout the training program.

OTHER OUTCOMES:
Time to pulmonary exacerbation | 12 Months
  The average time to exacerbation between groups will be analysed post trial.

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Teschler, Prof. Dr. med., Principal Investigator — Dept. Respiratory & Sleep Medicine - Ruhrlandklinik
Locations (1):
- Ruhrlandklinik, Tuschen, Hesse, Germany